CLINICAL TRIAL: NCT03305887
Title: A Prospective, Multicenter, Randomized Controlled Study to Evaluate the Wound Closure Efficiency of STRATAFIX™ Symmetric PDS™ Plus Knotless Tissue Control Device Compared to Conventional Sutures in Total Knee Arthroplasty (TKA)
Brief Title: Symmetric on Total Knee Arthroplasty (TKA)
Acronym: SFX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Medical, China (Industry)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); China-Japan Union Hospital, Jilin University (Other); Nanfang Hospital, Southern Medical University (Other); Tongji Hospital (Other); Chinese PLA General Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESC-16-001
Record Dates: First submitted 2017-01-13; First posted 2017-10-10 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Wound Closure
Keywords: TKA; Barbed suture; Surgical time

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Barbed suture group (Experimental): The deep layer and the intermediate layer will be repaired and closed by using one "STRATAFIX™ Symmetric" Knotless Tissue suture respectively. STRATAFIX Spiral sutures will be used to close the intradermal layer and the DERMABOND™ Advance™ Skin Closure System, a topical skin adhesive (TSA) will be applied to the skin surface to tissue approximation.
  Interventions: Device: "STRATAFIX™ Symmetric" Knotless Tissue; Device: "STRATAFIX Spiral" sutures; Device: DERMABOND™ Advance™ Skin Closure System
- Conventional suture group (Active Comparator): VICRYL® Plus sutures will be used to close the deep and the intermediate layers with interrupted suturing manner. STRATAFIX Spiral sutures will be used to close the intradermal layer and the DERMABOND™ Advance™ Skin Closure System, a topical skin adhesive (TSA) will be applied to the skin surface to tissue approximation.
  Interventions: Device: VICRYL® PLUS; Device: "STRATAFIX Spiral" sutures; Device: DERMABOND™ Advance™ Skin Closure System

INTERVENTIONS:
Device: "STRATAFIX™ Symmetric" Knotless Tissue — This devices will be used in deep and intermediate layers of barbed suture group.
  Other Names: STRATAFIX Symmetric
  Arms: Barbed suture group
Device: VICRYL® PLUS — This devices will be used in deep and intermediate layers of conventional suture group.
  Other Names: Polyglactin 910
  Arms: Conventional suture group
Device: "STRATAFIX Spiral" sutures — This devices will be used in intradermal layer of both barbed suture and conventional suture group.
  Other Names: Spiral
Device: DERMABOND™ Advance™ Skin Closure System — This devices will be used in skin layer of both barbed suture and conventional suture group.
  Other Names: DERMABOND

SUMMARY:
A post-marketing prospective, multicenter, randomized controlled study to evaluate the wound closure efficiency of STRATAFIX™ Symmetric PDS™ Plus Knotless Tissue Control Device (STRATAFIX Symmetric PDS Plus) compared to conventional sutures in total knee arthroplasty (TKA)

DETAILED DESCRIPTION:
The primary objective of this prospective, randomized controlled study is to evaluate the wound closure efficiency of STRATAFIX Symmetric PDS Plus compared to conventional sutures in patients undergoing TKA. For the purpose of this study, wound closure efficiency is defined as the total time required to close the surgical incisions in patients undergoing TKA procedures using STRATAFIX Symmetric PDS Plus compared to those using traditional sutures. Secondary objectives will include the evaluation of differences in overall surgical procedure time, operating room (OR) time, length of stay, procedure costs, quality of life measures including pain, and range of motion (ROM). In addition, the difference in the safety profiles for both wound closure procedures will be evaluated through the analysis of the incidence of wound complications including dehiscence, wound infections, and other adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years and < 80 years of age;
2. Patient with osteoarthritis is scheduled to undergo elective unilateral TKA;
3. Patient is willing to participate in the study, comply with study requirements, follow-up schedule, and give written informed consent; and
4. Patient agrees not to schedule any additional elective surgical procedures until participation in this study is complete.

Exclusion Criteria:

1. Female patient who is pregnant or lactating at the time of screening;
2. Patient has a Body Mass Index (BMI) > 40 kg/m2;
3. Patient is not able to walk independently (inability to walk at least 10 consecutive meters without a walking aid);
4. Patient has had a surgical intervention during the past 30 days for treatment of painful joint or its underlying etiology;
5. Patient has had previous open surgeries on the affected joint other than arthroscopy;
6. Patient has active infectious collagen diseases (i.e. scleroderma) or any other condition that would interfere with wound healing;
7. Patient is allergic to poly (p-dioxanone), triclosan (IRGACARE®* MP) or D&C Violet No. 2;
8. Patient has diabetes with poor control, defined as fasting plasma glucose (FPG) ≥ 10.0 mmol/L;
9. Patient has a history of immunosuppressive drug use, including steroids, within the last 6 months;
10. Patient has undergone chemotherapy or radiation within the last 6 months prior to study enrollment or is scheduled to do so during the study period;
11. Patient has known personal or family history of keloid formation or hypertrophy;
12. Patient has other dermatologic conditions known to impair wound healing;
13. Patient is participating in any other investigational drug (within 30 days or 5 half-lives of an investigational drug) or device study;
14. Patient has any physical or psychological condition which would impair study participation; and
15. Patient is judged unsuitable for study participation by the investigator for any other reason.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patty Schleckser, Study Director — Ethicon, Inc.
Locations (7):
- China (7):
  - Chinese PLA general hospital, Beijing, Beijing Municipality
  - NanFang Hospital, Guangzhou, Guangdong
  - Tongji Hospital affiliated Tongji medical college huazhonguniversity of science&technology, Wuhan, Hubei
  - Jiangsu province hospital, Nanjing, Jiangsu
  - Jilin University Chinese Japanese Friendship Hospital, Changchun, Jilin
  - second affiliated hospital of Xi'an Jiaotong university, Xi’an, Shanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- STRATAFIX Symmetric PDS Plus: an antibacterial (polydioxanone) monofilament, synthetic absorbable device prepared from polydioxanone (p-dioxanone)
- Conventional Sutures: Conventional Sutures is VICRYL Plus(Polyglactin 910)
Period: Overall Study
Arm/Group | STRATAFIX Symmetric PDS Plus | Conventional Sutures
Started (First Patient In 2017.06.12) | 91 | 93
Completed (Last Patient Out 2018.05.21) | 80 | 83
Not Completed | 11 | 10

BASELINE CHARACTERISTICS:
Population: All efficacy endpoints will be summarized descriptively by treatment group. The continuous variables will be summarized descriptively by number of subjects, mean, standard deviation, minimum, and maximum. Categorical data will be summarized descriptively by frequencies along with the associated percentages.
Groups:
- Total: Total of all reporting groups
Arm/Group | STRATAFIX Symmetric PDS Plus | Conventional Sutures | Total
Number analyzed (Participants) | 91 | 93 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 30 | 65
  >=65 years | 56 | 63 | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 68 | 138
  Male | 21 | 25 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 91 | 93 | 184
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Suturing Time
Description: The total time required to close the surgical incisions between treatment groups.
Time Frame: During Surgery
Population: total 184 patients enrolled in this study, and 5 patients have no suture time, because they withdrawn from study before surgery or violated protocol, etc.
Measure: Mean (97.5% Confidence Interval); unit: minuts
Arm/Group | STRATAFIX Symmetric PDS Plus | Conventional Sutures
Number analyzed (Participants) | 90 | 89
minuts | 15.516 [3.083 to 30.200] | 20.864 [10.267 to 43.617]

ADVERSE EVENTS:
Time Frame: 42 days
Description: An Adverse Events (AE) is defined as any untoward medical occurrence, regardless of its relationship to the study device (study suture) or the study procedure (Total Knee Arthoplasty). An untoward medical occurrence includes any new, undesirable medical experience or worsening of a pre-existing condition, which occurs at any point from the surgery to Final Visit.
Groups:
- STRATAFIX Symmetric PDS Plus: an antibacterial (polydioxanone) monofilament, synthetic absorbable device prepared from polydioxanone (p-dioxanone) total 90 patients had been collected Adverse Events(AE) related data, and 1 patient has no data in this group.
- Conventional Sutures: Conventional Sutures is VICRYL Plus (Polyglactin 910) total 89 patients had been collected Adverse Events(AE) related data, and 4 patient has no AE data in Conventional Sutures group.
Arm/Group | STRATAFIX Symmetric PDS Plus | Conventional Sutures
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/89
Serious Adverse Events (participants affected / at risk) | 3/90 | 2/89
Other Adverse Events (participants affected / at risk) | 8/90 | 14/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STRATAFIX Symmetric PDS Plus (N=90) | Conventional Sutures (N=89)
Postoperative pain/postoperative exudation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Incision subcutaneous hemorrhage and Incision exudate (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
inflammatory reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Incision infection (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain after knee replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STRATAFIX Symmetric PDS Plus (N=90) | Conventional Sutures (N=89)
white blood cell increment (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
red blood cell decrement (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
monocytes increment (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
inflammatory reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Incision inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Limb swelling （left） (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hemorrhagic seepage of wound (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tension vesicle around the wound (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
seepage of wound (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hemorrhagic infiltration of wound (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemorrhagic seepage of wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
lower limb swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Contagious eczema rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
drug fever (Immune system disorders) | 0 (0) | 1 (1)
hypoalbuminemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the principal investigator(PI) is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT03305887/SAP_000.pdf
  • Study Protocol (2017-05-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT03305887/Prot_001.pdf